CLINICAL TRIAL: NCT04603859
Title: When to INDuce for OverWeight? - a Randomised Controlled Trial (WINDOW)
Brief Title: When to INDuce for OverWeight? (WINDOW)
Acronym: WINDOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Randers Regional Hospital (Other); Herning Hospital (Other); Central Jutland Regional Hospital (Other); Nykøbing Falster County Hospital (Other); Odense University Hospital (Other); Rigshospitalet Juliane Marie Centret (Unknown); Kolding Sygehus (Other); Herlev Hospital (Other); Hvidovre University Hospital (Other); North Zealand's Hospital (Unknown); Zealand University Hospital - Roskilde (Unknown)
Responsible Party: Principal Investigator, Lise Krogh, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WINDOW
Record Dates: First submitted 2020-10-12; First posted 2020-10-27 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy; Obesity; Parturition
Keywords: Induction of labor; Expectant management; Cesarean section
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elective induction of labour (Experimental): Elective induction of labour at 39 gestational weeks and 0 to 3 days.
  Interventions: Procedure: Elective induction of labor at 39 gestational weeks and 0 to 3 days
- Expectant management (No Intervention): Awaiting spontaneous labor.

INTERVENTIONS:
Procedure: Elective induction of labor at 39 gestational weeks and 0 to 3 days — Elective induction of labor (eIOL) according to local policies
  Other Names: eIOL
  Arms: Elective induction of labour

SUMMARY:
The rate of overweight and obese women becoming pregnant is increasing. Obesity in pregnancy along with delivery by cesarean section in obese women is associated with several complications as compared to normal weight women. The longer the woman is pregnant, the longer she is at risk. In an otherwise low-risk pregnant woman at term, it is an ongoing clinical dilemma, whether the benefits of elective induction of labor and termination of the pregnancy will outweigh the potential harms from concomitant induction and delivery process. The proposed study is a randomized controlled study of elective induction versus expectant management in obese women. The study will be carried out as a national multicenter study with inclusion of 1900 participants from Danish delivery wards. The null hypothesis is that the caesarean section rate is similar with elective induction of labor at 39 weeks of gestation, compared with expectant management among pregnant women with pre- or early pregnancy BMI≥30.

DETAILED DESCRIPTION:
Background The World Health Organization (WHO) defines overweight as a body mass index (BMI) of ≥25 kg/m2 and obesity as a BMI of ≥30 kg/m2. Overweight and obesity are rising dramatically worldwide. In fertile women, the prevalence of obesity is one third in the United States, 20% in the United Kingdom, and 12-13% in Denmark. The association between obesity in pregnancy and the risk of gestational complications increases with increasing BMI. Among other complications, obesity in pregnancy is associated with increased risk of caesarean delivery. Delivery by caesarean section further adds significant risks of wound infection or other infectious morbidity in obese women as compared to normal weight women. The longer the woman is pregnant, the longer the risk of pregnancy complications remains. In an otherwise low-risk pregnant woman at term, it is an on-going clinical dilemma, whether the benefits of elective induction of labor (eIOL) and termination of the pregnancy will outweigh the potential harms from the concomitant induction and delivery process. Regarding delivery complications, based on data from historical cohorts, eIOL has traditionally been associated with an increased risk of caesarean section and instrumental delivery. Therefore, expectant management has been the preferred clinical option. This interpretation has now been challenged by a randomized trial (ARRIVE) with >6000 low-risk pregnant women where eIOL at 39 weeks of gestation was associated with lower caesarean delivery rates. There are no randomized studies in obese women, but two larger observational studies did find lower odds of caesarean delivery in obese women with eIOL as compared to awaiting labor onset. Hence, a randomized trial that would compare caesarean delivery among obese women whose labor is induced with those expectantly managed is warranted. The proposed study will provide new and important knowledge into the area of induction of labor among overweight and obese women with potential great international impact for the future raising number of pregnant women in this subgroup.

With this trial, the investigators aim to compare the risk of caesarean section in obese (BMI ≥ 30 kg/m2), but otherwise low-risk women with eIOL as compared to expectant management.

Materials and methods

The study is a multicenter randomized controlled trial with an allocation ratio of 1:1 in the two following arms:

* Intervention arm/elective induction of labor in pregnancy at 39 gestational week and 0 to 3 days: Induction is performed according to local policy for induction of labor.
* Comparison arm/expectant management: Waiting for spontaneous onset of labor unless a situation develops necessitating either induction of labor or caesarean section.

  1900 low-risk pregnant women with a pre- or early pregnancy BMI ≥ 30 carrying a singleton pregnancy will be recruited from the Danish delivery wards. In each trial site, a physician investigator will be responsible for the enrolment, the electronically randomization, and data collection.

The primary endpoint is the caesarean section rate. Among others there will be secondary endpoints on instrumental delivery, onset of labor, methods of induction, perinatal and postpartum complications both maternal and neonatal along with data on women's experience on birth measured by a questionnaire survey four to six weeks post-partum.

Ethics The study will be conducted in accordance with the ethical principles outlined in the latest version of the 'Declaration of Helsinki' and the 'Guideline for Good Clinical Practice' related to experiments on humans. The Central Denmark Region Committee on Biomedical Research Ethics, and The Danish Health Authorities have approved the study.

Perspectives In perspective, more than 39% of the world's population is overweight and 13% are obese by the WHO classification. Pregnant overweight women are at increased risk of pregnancy and delivery complications, and there is a need to improve maternity care for this subgroup of women. The results of this trial have the potential to generate important knowledge for the improvement of delivery in obese women and they will add key information to an on-going discussion of the effects of labor induction before term. Any possible harm or disadvantage to the individual study participant is outweighed by the possible benefit to the increasing number of obese women who will be pregnant in the future.

ELIGIBILITY:
Inclusion Criteria:

• Pregnant women with pre- or early pregnancy BMI ≥ 30 kg/m2

Exclusion Criteria:

* Legal or ethical considerations: maternal age <18 years, language difficulties requiring an interpreter or translator
* Multiple pregnancy
* Previous caesarean section
* Uncertain gestational age, defined as gestational age determined by other measurements than the Crown-Rump length (CRL) Measurement
* Planned elective caesarean section at time of randomisation
* Fetal contraindications to IOL at time of randomisation: e.g. non-cephalic presentation, or other fetal conditions contraindicating vaginal delivery
* Fetal contraindications to expectant management at time of randomisation
* Maternal contraindications to IOL at time of randomisation: e.g. placenta previa/accreta, vasa previa
* Maternal contraindications to expectant management at time of randomisation: e.g. maternal medical conditions, ultrasonically diagnosed oligohydramnios (DVP< 2 cm), signs of labour including pre-labour rupture of membranes (PROM)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Caesarean section | At delivery
  number (no.)

SECONDARY OUTCOMES:
Mode of delivery if not by caesarean | At delivery
  * Vaginal delivery - no.
  * Vaginal assisted delivery - no.
Mode of delivery | At delivery
  * Caesarean section - percent
  * Vaginal delivery - percent
  * Vaginal assisted delivery - percent
Vaginal assisted delivery | At delivery
  * Forceps - no.
  * Ventouse - no.
Indication for caesarean section (more than one indication is possible) | At delivery
  * Labour dystocia - no.
  * Fetal distress - no.
  * Maternal request - no.
  * Suspected macrosomia - no.
  * Non-cephalic presentation - no.
  * Extensive vaginal bleeding - no.
  * Suspected uterine rupture - no.
  * Maternal or fetal complication/condition (free text) - no.
  * Other indication for caesarean section (free text) - no.
Indication for vaginal assisted delivery (more than one is possible) | At delivery
  * Labour dystocia - no.
  * Fetal distress - no.
  * Maternal request - no.
  * Other indication for assisted vaginal delivery (free text) - no.
Use of epidural | At delivery
  no.
Damage to internal organs (bladder, bowel or ureters) | At delivery to 30 days postpartum
  no.
Uterine scar dehiscense or rupture | At delivery
  no.
Complications | At delivery
  * Minor shoulder dystocia defined as the need for McRobert's maneuver - no.
  * Major shoulder dystocia defined as the need for procedures other than McRobert's maneuver - no.
  * Clinical suspicion of abruption of the placenta leading to an intervention in labour - no.
  * Cord prolapse - no.
  * Maternal fever defined as temperature >38,2 / >38,0 degrees celsius with / without epidural - no.
  * Perineal 3rd degree laceration - no.
  * Perineal 4th degree laceration - no.
  * Episiotomy - no.
Postpartum haemorrhage | 0-2 hours postpartum
  * Blood loss >500ml - no.
  * Blood loss >1000ml - no.
  * Blood transfusion - no. Time Frame [0-2 days postpartum]
Hysterectomy | At delivery to 30 days postpartum
  no.
Postpartum morbidity | 0-30 days postpartum
  * Puerperal infection treated in hospital - no.
  * Other severe postpartum conditions treated in hospital (free text) - no.
Maternal admission to Intensive Care Unit | Enrollment to 30 days postpartum
  no.
Maternal cardiopulmonary arrest | Enrollment to 30 days postpartum
  no.
Maternal death | Enrollment to 30 days postpartum
  no.
Primary neonatal composite including any of the following; | Enrollment to 28 days of life
  * Perinatal death (stillbirth and neonatal)
  * The need for respiratory support if admitted to a neonatal department (intubation and mechanical ventilation, oxygen, continuous positive airway pressure (CPAP), or high-flow nasal cannula (HNFC)). Time Frame [within 72 hours after birth]
  * Apgar score < 4 at 5 minutes
  * Hypoxic-ischemic encephalopathy (defined as the need for therapeutic hypothermia)
  * Seizures
  * Infection (defined as antibiotic treatment continuously for 7 days minimum)
  * Meconium aspiration syndrome
  * Birth trauma (bone fracture, Duchenne-Erbs palsy, or retinal hemorrhage)
  * Intracranial or subgaleal hemorrhage
  * Hypotension requiring vasopressor support
Components of the primary neonatal composite will additionally be reported separately | Enrollment to 28 days of life
  * Perinatal death (stillbirth and neonatal) - no.
  * The need for respiratory support if admitted to a neonatal department (intubation and mechanical ventilation, oxygen, continuous positive airway pressure (CPAP), or high-flow nasal cannula (HNFC)). Time Frame [within 72 hours after birth] - no.
  * Apgar score < 4 at 5 minutes - no.
  * Hypoxic-ischemic encephalopathy (defined as the need for therapeutic hypothermia) - no.
  * Seizures - no.
  * Infection (defined as antibiotic treatment continuously for 7 days minimum) - no.
  * Meconium aspiration syndrome - no.
  * Birth trauma (bone fracture, Duchenne-Erbs palsy, or retinal hemorrhage) - no.
  * Intracranial or subgaleal hemorrhage - no.
  * Hypotension requiring vasopressor support - no.
Neonatal trauma composite including any of the following; | At delivery to 28 days of life
  * Birth trauma (bone fracture, Duchenne-Erbs palsy, or retinal hemorrhage)
  * Intracranial or subgaleal hemorrhage
Neonatal asphyxia composite including any of the following; | At delivery to 28 days of life
  * Apgar score < 4 at 5 minutes
  * Umbilical cord pH-value < 7.0 (allow missing data)
  * Umbilical cord standard base excess (sBE) < -15.0 mmol/l (allow missing data)
  * Seizures
  * Hypoxic-ischemic encephalopathy (defined as the need for therapeutic hypothermia)
Apgar score at 5 minutes | 5 minutes of life
  * Apgar score <4 - no.
  * Apgar score of 4-7 - no.
Umbilical cord arterial and venous blood sample (allow missing data) | 0-30 minutes of life
  * pH-value < 7.0 - no.
  * sBE < -15.0 mmol/l - no.
Neonatal admission | 0-72 hours of life
  no.
Respiratory support during neonatal admission | 0-28 days of life
  * CPAP (y/n) - no.
  * HNFC (y/n) - no.
  * Oxygen supplement treatment (y/n) - no.
  * Ventilator treatment (y/n) - no.
Other treatment during neonatal admission | 0-28 days of life
  * Therapeutic hypothermia (y/n) - no.
  * Vasopressor support (y/n) - no.
  * Antibiotic treatment continuously for 7 days minimum (y/n) - no.

OTHER OUTCOMES:
Neonatal characteristics 1 | At delivery
  * Female sex - no.
  * Birth weight > 4500 grams (y/n) - no.
Neonatal characteristics 2 | At delivery
  - Mean birth weight - grams
Maternal experience on birth | 4-6 weeks postpartum
  Childbirth Experience Questionnaire Scoring range is 1 to 4 where higher ratings reflect more positive experiences
Maternal postnatal depression | 4-6 weeks postpartum
  * Major Depression Inventory (MDI)
  * Edinburgh Postnatal Depression Score Scoring range is 1 to 4 where higher ratings reflect more positive experiences

CONTACTS AND LOCATIONS:
Overall Officials: Lise Q Krogh, MD, Principal Investigator — Aarhus University Hospital; Julie Glavind, MD, PhD, Study Chair — Aarhus University Hospital; Sidsel Boie, MD, PhD, Study Chair — Randers Regional Hospital; Jens Fuglsang, MD, PhD, Study Chair — Aarhus University Hospital; Tine B Henriksen, MD, PhD, Study Chair — Aarhus University Hospital; Jim Thornton, MD, PhD, Study Chair — Nottingham University; Katja A Taastrøm, Midwife, MSc, Study Chair — Aarhus University Hospital; Anne Cathrine M Kjeldsen, Midwife, MSc, Study Chair — Aarhus University Hospital
Locations (12):
- Denmark (12):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Juliane Marie Centre, Copenhagen
  - Herlev Hospital, Herlev
  - Gødstrup Regional Hospital, Herning
  - North Zealand's Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Kolding Hospital, Kolding
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Zealand University Hospital, Roskilde
  - Viborg Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be publicly available in an anonymised form using an open data repository (i.e. CERN) or another equivalent database.
  All relevant trial-related documents will be shared along with the data.
Time Frame: Beginning three months and ending three years after the publication of the last trial results.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee. Interested parties will be able to request the data by contacting the trial sponsor. Authorship of publications emerging from the shared data will follow standard authorship guidelines and will include authors from the WINDOW study group depending on the nature of their involvement.

REFERENCES:
- [Derived] Krogh LQ, Boie S, Henriksen TB, Thornton J, Fuglsang J, Glavind J. Induction of labour at 39 weeks versus expectant management in low-risk obese women: study protocol for a randomised controlled study. BMJ Open. 2022 Apr 25;12(4):e057688. doi: 10.1136/bmjopen-2021-057688. PMID 35470194

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol including Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04603859/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed Statistical Analysis Plan (separate) (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT04603859/SAP_001.pdf